CLINICAL TRIAL: NCT00443040
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating Asimadoline on the Duration of POI in Subjects Undergoing Laparoscopic/Hand-Assisted Lap Segmental Colonic Resection Secondary to Colon Cancer, Polypectomy or Diverticulitis
Brief Title: Asimadoline for the Treatment of Post-Operative Ileus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor enrollment (31 of a planned 114 subjects were randomized and evaluable)
Sponsor: Tioga Pharmaceuticals (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASMP2004
Record Dates: First submitted 2007-02-27; First posted 2007-03-05 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2011-11

CONDITIONS: Post-Operative Ileus
MeSH Terms: interventions — asimadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Asimadoline 1.0 mg (Active Comparator): Asimadoline 1.0 mg b.i.d.
  Interventions: Drug: Asimadoline
- Asimadoline 3.0 mg (Active Comparator): Asimadoline 3.0 mg b.i.d.
  Interventions: Drug: Asimadoline

INTERVENTIONS:
Drug: Asimadoline — Asimadoline was provided in coated tablets of 1.0 mg strength. Subjects were given 3 tablets of study drug 90 minutes prior to their operation and then 3 tablets b.i.d. for up to 10 post-operative doses. Subjects randomized to receive 3.0 mg of asimadoline received three 1.0 mg asimadoline tablets at each scheduled dose, while those randomized to receive 1.0 mg of asimadoline received two placebo tablets and one 1.0 mg asimadoline tablet at each scheduled dose.
  Other Names: EMD 61 753; EMR 63 320
  Arms: Asimadoline 1.0 mg; Asimadoline 3.0 mg
Drug: Placebo — Placebo was provided in coated tablets identical in appearance to asimadoline tablets. Subjects were given 3 tablets of placebo 90 minutes prior to their operation and then 3 placebo tablets b.i.d. for up to 10 post-operative doses.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of asimadoline in patients who have undergone a laparoscopic segmental colectomy and determine whether it reduces the time to recovery of bowel function compared to placebo.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study was designed to evaluate the efficacy and tolerability of two dose levels of asimadoline on the duration of post-operative ileus in subjects undergoing laparoscopic or hand-assisted laparoscopic colon resections. Subjects meeting entry criteria were randomized in a 1:1:1 ratio to receive either asimadoline 1.0 mg, asimadoline 3.0 mg or a placebo. One hundred and fourteen subjects were planned, and in the event that a subject was converted from a laparoscopic surgery to an open surgery (laparotomy), that subject would be discontinued from the trial and followed for safety only. The protocol allowed subjects converted to open procedures to be replaced. The first dose was administered approximately 90 minutes pre-operatively, and subsequent dosing was b.i.d. for up to 10 post-operative doses. Subjects were dosed with study drug only while in the hospital. After discharge, they were followed for an additional 28 days. Total study duration for each patient was approximately 5 to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-80
* Must be scheduled to undergo a laparoscopic/hand-assisted laparoscopic segmental colectomy
* Must sign an ICF
* Females of childbearing potential must have a negative pregnancy test at screening

Exclusion Criteria:

* Subjects with evidence of a biochemical or structural abnormality of the GI tract or other co-morbid illness that may impact the ability to interpret the safety and efficacy data
* Pregnant or breastfeeding females
* Use of investigational drugs in previous 30 days
* Refusal to discontinue prohibited concomitant medications
* Chronic use of prescription narcotics over the previous 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Mangel, MD, PhD, Study Chair — CMO
Locations (4):
- United States (4):
  - Lahey Clinic, Burlington, Massachusetts
  - Washington University, St Louis, Missouri
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Marks Colorectal Surgical Associates, Wynnewood, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Asimadoline 1.0 mg | Asimadoline 3.0 mg | Placebo
Started | 14 | 11 | 10
Completed | 10 | 11 | 9
Not Completed | 4 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Converted to an open laparotomy | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asimadoline 1.0 mg | Asimadoline 3.0 mg | Placebo | Total
Number analyzed (Participants) | 14 | 11 | 10 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 6 | 22
  >=65 years | 4 | 5 | 4 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (9.7) | 60 (12.9) | 57 (15.3) | 58 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 3 | 15
  Male | 9 | 4 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 14 | 11 | 10 | 35

OUTCOME MEASURES:

1. Secondary Outcome: Time to Tolerating Solid Food
Description: Time to tolerating solid food (toleration is defined as the absence of nausea or vomiting) within 4 hours of ingesting a meal
Time Frame: 4 hours of ingesting a meal
Reporting Status: Not Posted
Measure: Number; unit: participants

2. Secondary Outcome: Time to First Passage of Flatus
Time Frame: Daily for 38 days
Reporting Status: Not Posted
Measure: Number; unit: participants

3. Secondary Outcome: Time to First Bowel Movement
Time Frame: Daily for 38 days
Reporting Status: Not Posted
Measure: Number; unit: participants

4. Secondary Outcome: Time to Writing of Hospital Discharge Order
Time Frame: Daily for 38 days
Reporting Status: Not Posted
Measure: Number; unit: participants

5. Secondary Outcome: Nausea Score
Time Frame: Daily for 38 days
Reporting Status: Not Posted

6. Secondary Outcome: Vomiting Score
Time Frame: Daily for 38 days
Reporting Status: Not Posted

7. Secondary Outcome: Pain Score
Time Frame: Daily for 38 days
Reporting Status: Not Posted

8. Primary Outcome: Time to Return of Upper and Lower GI Function
Description: The time to first bowel movement or the time to tolerating solid food, whichever occurs later.
Time Frame: Daily for 38 days
Population: As the study was terminated early due to poor enrollment (31 of a planned 114 subjects were randomized and evaluable), no formal efficacy analyses were conducted.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Asimadoline 1.0 mg | Asimadoline 3.0 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Nasogastric Tube Re-insertion
Description: Proportion of subjects with nasogastric tube re-insertion
Time Frame: Daily for 38 days
Reporting Status: Not Posted

10. Secondary Outcome: Post-operative Analgesic Use
Time Frame: Daily for 38 days
Reporting Status: Not Posted

11. Secondary Outcome: Adverse Events
Description: Adverse events grouped by body system
Time Frame: Daily for 38 days
Reporting Status: Not Posted

12. Secondary Outcome: Laboratory Values
Description: Changes in laboratory values.
Time Frame: Daily for 38 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Asimadoline 1.0 mg | Asimadoline 3.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/11 | 1/10
Other Adverse Events (participants affected / at risk) | 14/14 | 11/11 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asimadoline 1.0 mg (N=14) | Asimadoline 3.0 mg (N=11) | Placebo (N=10)
bleeding gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
omental necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asimadoline 1.0 mg (N=14) | Asimadoline 3.0 mg (N=11) | Placebo (N=10)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7) | 4 (4)
Procedural Pain (Injury, poisoning and procedural complications) | 4 (4) | 5 (5) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Potassium Decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Painful defaecation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal functional disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Suprapubic pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; no efficacy analysis was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator understands and agrees that the first publication of the results of the Research Study, if any, shall be a multicenter publication of the results from all sites. Institution shall not publish, present, or use any results of the Research Study for any purpose until such Research Study has been completed in its entirety at all sites and until such multi-center study publication has been published or for a period of one year following such completion, whichever occurs first.